CLINICAL TRIAL: NCT04807387
Title: Newly-designed Vaginal Stent to Improve Tissue Healing for Girls and Women With Congenital and Reproductive Anomalies
Brief Title: Newly Designed Vaginal Stent to Improve Patient Comfort and Healing Following Vaginal Surgery or Vaginal Radiation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After enrolling 6 healthy participants the study is being put on halted due to funding and personnel gap. All participants have been informed, per study IRB, of study status.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); BioTex, Inc. (Industry)
Responsible Party: Principal Investigator, Julie Hakim, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45549; 5R44HD092156-03 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-19 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Vaginal Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Healthy participants: acute (Experimental): Healthy participants will wear one of two vaginal stents for 24 hours, followed by a 24 hour wash out period. They will then wear the second vaginal stent for 24 hours. After both stents have been worn, the participants will choose the most comfortable stent.
  Interventions: Device: Vaginal Stent A; Device: Vaginal Stent B
- Healthy participants: chronic (Experimental): Healthy participants will wear the stent chosen to be the more comfortable for 2 weeks without removal.
  Interventions: Device: Vaginal Stent
- Pediatric participants: post vaginal surgery (Experimental): Pediatric participants will wear the vaginal stent for 2 weeks after undergoing vaginal surgery.
  Interventions: Device: Vaginal Stent
- Adult participants: post vaginal brachytherapy (Experimental): Adult participants undergoing vaginal brachytherapy for cancer treatment will wear the stent for 2 weeks, be evaluated by a physician, and wear the stent for an additional 2 weeks.
  Interventions: Device: Vaginal Stent

INTERVENTIONS:
Device: Vaginal Stent A — Ring stent
  Arms: Healthy participants: acute
Device: Vaginal Stent B — Flower stent
  Arms: Healthy participants: acute
Device: Vaginal Stent — Vaginal stent chosen from A or B that is the most comfortable
  Arms: Adult participants: post vaginal brachytherapy; Healthy participants: chronic; Pediatric participants: post vaginal surgery

SUMMARY:
Each year, females need surgery to create a vaginal canal or pelvic radiation to treat cancer. The result is often a narrowing or scarring of their vagina. To aid in healing a stent is often placed. However, current stents are poorly designed. The goal of this trial is to test newly designed vaginal stents, with the hope of replacing the poorly retained and uncomfortable standard of care. This trial has two aims. In the first aim, healthy participants will evaluate two newly designed vaginal stents for retention, comfort, and safety over 24 hours. The preferred stent will then be worn by the healthy participants for 2 weeks, again evaluating retention, comfort, and safety. In the second aim, the stents will be evaluated by two different patient populations. Adolescent participants undergoing vaginal surgery for genetic anomalies, will have a stent placed following surgery for continuous wear for 2 weeks. Adult participants undergoing vaginal brachytherapy will have the stent placed following the final brachytherapy treatment. These participants will wear the stent continuously for 2 weeks, followed by an additional 2 weeks of continuous wear. Each participant will evaluate the stent for retention, comfort, and safety. We hypothesize the newly designed stents will be retained longer and be more comfortable compared to current standards of care.

DETAILED DESCRIPTION:
After surgery or radiation to the vaginal area, a common patient risk is that their vaginal tissue sticks together and scars. This can cause the vaginal canal to narrow or shorten. This can occur in up to 73% of patients and to fix the scarring, more surgery or uncomfortable procedures may be needed to widen the canal. To prevent the problem of scarring after surgery or radiation, patients should wear a stent to hold open the vaginal canal. Unfortunately, the current stents are poorly made and not very advanced. The result can be a poor fit to the vagina, movement of the stent, and patients not being able to wear the stent for a long enough time to keep the vaginal tissue from scarring.

The first aim of this trial is for healthy participants to evaluate two newly designed stents. Each participant will have a stent placed for 24 hours, removed for 24 hours, and the second stent placed for 24 hours. The participants will evaluate the stent on comfort (during insertion, wearing, and removal), retention, any impact on daily functions, and chose which stent performed better overall. That stent will then be placed in the healthy participants for 2 weeks of continuous wear. Participants will answer daily questionnaires on comfort, retention, and any adverse effects. Physicians will also be asked to complete questionnaires at each appointment related to stent performance.

The second aim of the trial is for two different patient populations to evaluate the preferred stent chosen by the healthy participants. Adolescent girls undergoing vaginal reconstructive surgery for vaginal anomalies will have a stent placed following surgery. During the two weeks of continuous wear, participants will be asked to answer daily questionnaires on comfort, retention, and adverse effects. The stent will be removed at two weeks, and participants will be asked to complete a follow-up questionnaire at each of their standard of care appointments, 2, 4, and 6 weeks, 3, 6, and 12 months. Adult females undergoing vaginal brachytherapy will have a stent placed after their last brachytherapy treatment. The participants will wear the stent continuously for 2 weeks and be asked to answer daily questionnaires on comfort, retention, and adverse effects. Participants will have a 2-week follow-up, during which the stent will be removed, they will be examined, and the stent will be replaced for 2 more weeks of continuous wear. At the 4-week follow-up, the stent will be removed and subsequent standard of care follow-ups will continue at 3, 6, and 12 months. Physicians will also be asked to complete questionnaires at each appointment related to stent performance.

During all phases of the trial, the data safety monitoring board will meet at regularly scheduled meetings and immediately after any severe or unanticipated adverse event. After our 12 months of follow up, data collected from both participant and physician questionnaires will be analyzed by the study bio-statistician and compared to retrospective data.

ELIGIBILITY:
Inclusion Criteria (healthy participants):

* Not pregnant
* participant consent or parent/guardian consent & participant assent
* Understand requirements of study
* Agree to abide by study restrictions
* Able to travel to Houston
* Understand English or Spanish to a 5th grade level
* No prior history of vaginal surgery or radiation

Inclusion Criteria (pediatric participants):

* Not pregnant
* participant consent or parent/guardian consent & participant assent
* Understand requirements of study
* Agree to abide by study restrictions
* Able to travel to Houston
* Understand English or Spanish to a 5th grade level
* Undergoing vaginal surgery

Inclusion Criteria (adult radiation participants):

* Not pregnant
* participant consent or parent/guardian consent & participant assent
* Understand requirements of study
* Agree to abide by study restrictions
* Able to travel to Houston
* Understand English or Spanish to a 5th grade level
* Undergoing vaginal brachytherapy

Exclusion Criteria (all arms):

* Non-English or Spanish speaker
* Pregnant
* BMI > 45
* Diabetic neuropathy limiting use of hands
* Other limited mobility of hands
* Vaginismus
* Urinary retention
* Vaginal bacterial infection
* Vaginal fungal infection
* Allergies to stent materials
* Seizure disorder
* Pain with sexual intercourse or tampon insertion

Ages: 13 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie CE Hakim, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ring Stent First, Then Flower Stent: Healthy participants will wear one of two vaginal stents for 24 hours, followed by a 24 hour wash out period. They will then wear the second vaginal stent for 24 hours. After both stents have been worn, the participants will choose the most comfortable stent.
  Vaginal Stent A: Ring stent
  Vaginal Stent B: Flower stent
- Flower Stent First, Then Ring Stent: Healthy participants will wear one of two vaginal stents for 24 hours, followed by a 24 hour wash out period. They will then wear the second vaginal stent for 24 hours. After both stents have been worn, the participants will choose the most comfortable stent.
  Vaginal Stent B: Flower stent
Period: Overall Study
Arm/Group | Ring Stent First, Then Flower Stent | Flower Stent First, Then Ring Stent
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Participants: Acute
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Vaginal Stent as Comfortable.
Description: Participants will report daily on stent comfort and any disruption to normal daily activities.
Time Frame: 24 hours from stent placement
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Participants: Acute - Vaginal Stent A: Ring Stent: Healthy participants will wear one of two vaginal stents for 24 hours, followed by a 24 hour wash out period. They will then wear the second vaginal stent for 24 hours. After both stents have been worn, the participants will choose the most comfortable stent.
  Vaginal Stent A: Ring stent
- Healthy Participants: Acute - Vaginal Stent B: Flower Stent: Healthy participants will wear one of two vaginal stents for 24 hours, followed by a 24 hour wash out period. They will then wear the second vaginal stent for 24 hours. After both stents have been worn, the participants will choose the most comfortable stent.
  Vaginal Stent B: Flower stent
Arm/Group | Healthy Participants: Acute - Vaginal Stent A: Ring Stent | Healthy Participants: Acute - Vaginal Stent B: Flower Stent
Number analyzed (Participants) | 4 | 5
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Through study completion (total 4 days)
Arm/Group | Healthy Participants: Acute - Vaginal Stent A: Ring Stent | Healthy Participants: Acute - Vaginal Stent B: Flower Stent
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04807387/Prot_SAP_000.pdf